CLINICAL TRIAL: NCT01373814
Title: Nutritional Therapy for Diabetic Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 10-1163
Record Dates: First submitted 2011-06-13; First posted 2011-06-15 (Estimated); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: T2DM (Type 2 Diabetes Mellitus)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this study is to determine if nutritional therapy can effectively treat/prevent T2DM and its consequent cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be >30 and <65 years of age, in order to limit the confounding affect of age on our endpoints.
* Subjects must have an ejection fraction >45% (based on their echocardiogram)
* Patients with T2DM and nonalcoholic fatty liver disease or steatohepatitis may be included since they have extensive evidence of steatosis.

Exclusion Criteria:

* Subjects who have had a myocardial infarction or resting ischemia (by history or as evidenced by hypo/akinesis on the pre-intervention echocardiogram) will be excluded because hypo/akinesis would affect our endpoints of LV mass and diastolic function.
* Subjects who are unstable, not able to lie flat for the imaging studies, unable to give informed consent, pregnant, lactating, with atrial fibrillation (which would compromise measurement of E'), or current smokers will be excluded.
* Subjects with other major systemic diseases per their clinical charts, history, physical exam, or significant renal insufficiency will also be excluded, as these other system diseases may affect our study endpoints and subject follow-up.
* We will exclude patients with significant LV systolic dysfunction (ejection fraction <45%)
* We will not exclude patients with sleep apnea because it does not detrimentally affect LV diastolic function.
* Subjects will be excluded a priori if they have any history or evidence of liver disease other than NAFLD, consumed >20 g alcohol per day.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known T2DM and who are not taking exogenous insulin.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2010-09-03; Primary Completion 2011-06-17 (Actual); Study Completion 2011-06-17 (Actual)

PRIMARY OUTCOMES:
cardiac function | 2 weeks
  cardiac function as measured by echocardiography incl. tissue Doppler

SECONDARY OUTCOMES:
liver steatosis | 2 weeks
  liver fat content as measured using MR spectroscopy
myocardial steatosis | 2 weeks
  fat in heart muscle as measured using MR spectroscopy
lipidomics | 2 weeks
  mass spectroscopy measures of plasma lipid species

CONTACTS AND LOCATIONS:
Overall Officials: Linda R Peterson, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Airhart S, Cade WT, Jiang H, Coggan AR, Racette SB, Korenblat K, Spearie CA, Waller S, O'Connor R, Bashir A, Ory DS, Schaffer JE, Novak E, Farmer M, Waggoner AD, Davila-Roman VG, Javidan-Nejad C, Peterson LR. A Diet Rich in Medium-Chain Fatty Acids Improves Systolic Function and Alters the Lipidomic Profile in Patients With Type 2 Diabetes: A Pilot Study. J Clin Endocrinol Metab. 2016 Feb;101(2):504-12. doi: 10.1210/jc.2015-3292. Epub 2015 Dec 10. PMID 26652763